CLINICAL TRIAL: NCT01493479
Title: Phase II Study of Fractionated 90Y Ibritumomab Tiuxetan (Zevalin)
Brief Title: Phase II Study of Fractionated 90Y Ibritumomab Tiuxetan (Zevalin) Radioimmunotherapy as an Initial Therapy of Follicular Lymphoma
Acronym: FIZZ
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Emmie Taylor, Lead Clinical Trial Manager, The Christie NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06_DOG05_33
Record Dates: First submitted 2011-12-14; First posted 2011-12-16 (Estimated); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — ibritumomab tiuxetan; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fractionated Initial Zevalin (Experimental)
  Interventions: Drug: 90Y Ibritumomab tiuxetan; Drug: Rituximab

INTERVENTIONS:
Drug: 90Y Ibritumomab tiuxetan — 2 x iv infusions of 11.1 MBq/kg. 1st infusion at week 1, 2nd during weeks 9-13. 2nd infusion may be reduced to 7.4MBq/kg in the case of grade 3 haematological toxicity following the 1st infusion.
  Other Names: Zevalin
Drug: Rituximab — All patients receive 2 x iv infusions of 250 mg/m2 Rituximab given 7-8 days apart prior to each zevalin infusion. The 2nd rituximab infusion is given immediately prior to Zevalin.
  In addition patients with greater than 20% bone marrow involvement at screening receive rituximab pretreatment prior to entering the main treatment phase of the trial, consisting of 4 x weekly iv doses of rituximab(375 mg/m2). This is followed by a repeat bone marrow biopsy, bone marrow involvement must have fallen to <= 20% to enter the main treatment phase of the trial.
  Other Names: Mabthera

SUMMARY:
90Y Ibritumomab tiuxetan (zevalin) has demonstrated consistently high response rates in patients who have received previous treatment for lymphoma. More than two-thirds of the patients who achieve CR go on to experience durable remissions lasting for years. Despite these highly promising clinical results with radioimmunotherapy (RIT) in relapsed follicular lymphoma there is very little data using RIT in previously untreated follicular lymphoma. The objective of this trial is to evaluate the safety and efficacy of two fractions of Zevalin in patients with previously untreated follicular lymphoma in a Phase II study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed CD20 +ve follicular lymphoma grades I to IIIa.
* Patients with at least one of the following symptoms requiring initiation of treatment: (as outlined by the modified BNLI/GELF criteria below)

  * Nodal mass > 7cm in its greater diameter
  * B symptoms
  * Elevated serum LDH or beta2-microglobulin
  * involvement of at least 3 nodal sites (each with a diameter > 3 cm)
  * symptomatic splenic enlargement
  * compressive syndrome
* Patients must have an ECOG performance status less than or equal to 2 and an anticipated survival of at least 6 months.
* Patients must have an absolute granulocyte count of above 1,500/mm3, and a platelet count of above 100,000/mm3 post 4 weeks of unlabelled Rituximab. A hemoglobin >= 8.0 g/dl
* Patients must have adequate renal function (defined as calculated creatinine clearance > 30 ml/mn), hepatic function (defined as total bilirubin <1.5 times upper limit of normal), and hepatic transaminases (defined as AST <5 times upper limit of normal)
* Patients must have given informed consent prior to study entry.

Exclusion Criteria:

* Patients with a mean of >20% of the intratrabecular marrow space involved with lymphoma on bone marrow biopsy following induction Rituximab therapy.
* Transformed follicular lymphoma and discordant lymphoma
* Patients with active obstructive hydronephrosis.
* Patients with initial disease bulk greater than 10cm.
* Patients with evidence of active infection requiring i.v. antibiotics at the time of study entry.
* Patients with congestive heart failure stage III or IV of NYHA classification, myocardial infraction or unstable angina within 6 months or other serious illness that would preclude evaluation.
* Patients with left VEF < 40%
* Patients with large pleural or peritoneal effusions.
* Patients with known HIV infection or active HBV (HbsAg positivity) or HCV infection.
* Known Hypersensitivity to murine antibodies or proteins
* Patients who are pregnant or breast-feeding. Male and female patients must agree to use effective contraception for 12 months following 90Y-ibritumomab tiuxetan antibody therapy.
* Patients with prior malignancy other than lymphoma, except for adequately-treated skin cancer, cervical cancer in situ, or other cancer for which the patient has been disease-free for 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2007-06-06 (Actual); Primary Completion 2011-01 (Actual); Study Completion 2015-11-06 (Actual)

PRIMARY OUTCOMES:
Overall response rate | Assessed 3 months post treatment
  According to Cheson criteria to standardize response for non-Hodgkin's lymphoma, 1999.
Combined Complete Response rate | Assessed 3 months post treatment
  According to Cheson criteria to standardize response for non-Hodgkin's lymphoma, 1999.
Partial Response Rate | Assessed 3 months post treatment
  According to Cheson criteria to standardize response for non-Hodgkin's lymphoma, 1999.

SECONDARY OUTCOMES:
Time to disease progression | Assessed 3 months post treatment, repeated assessment up to 5 years follow-up
Response duration | Assessed 3 months post treatment, repeated assessment up to 5 years follow-up
  To be assessed for patients achieving a response, including assessment of overall survival and time until next treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Illidge, Prof, Principal Investigator — The Christie NHS Foundation Trust
Locations (7):
- France (3):
  - Centre Hospitalier Universitaire de Lille, Lille
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Centre Henri Becquerel, Rouen
- United Kingdom (4):
  - St George's Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - Poole Hospital NHS Foundation Trust, Poole
  - Southampton University Hospital, Southampton

REFERENCES:
- [Derived] Illidge TM, Mayes S, Pettengell R, Bates AT, Bayne M, Radford JA, Ryder WD, Le Gouill S, Jardin F, Tipping J, Zivanovic M, Kraeber-Bodere F, Bardies M, Bodet-Milin C, Malek E, Huglo D, Morschhauser F. Fractionated (9)(0)Y-ibritumomab tiuxetan radioimmunotherapy as an initial therapy of follicular lymphoma: an international phase II study in patients requiring treatment according to GELF/BNLI criteria. J Clin Oncol. 2014 Jan 20;32(3):212-8. doi: 10.1200/JCO.2013.50.3110. Epub 2013 Dec 2. PMID 24297953